CLINICAL TRIAL: NCT00203177
Title: A Bi-national, Multicenter, Double-Blind, Randomized Study to Evaluate the Safety and Tolerability of Rasagiline Mesylate in Advanced Parkinson's Disease (PD) Patients With Motor Fluctuations Treated With Chronic Levodopa/Carbidopa Therapy.
Brief Title: Rasagiline in Advanced Parkinson's Disease Patients With Motor Fluctuations Treated With Levodopa/Carbidopa Therapy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Siyu Liu, MD, PhD, VP IR&D, Head of Global Clinical Operations, Teva Branded Pharmaceutical Products IR&D
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TVP - 1012/135 Double Blind
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-03

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental 1 (Experimental): 0.5 mg rasagiline mesylate oral once daily
  Interventions: Drug: rasagiline mesylate
- Expermental 2 (Experimental): 1.0 mg rasagiline mesylate oral once daily
  Interventions: Drug: rasagiline mesylate 1.0 mg

INTERVENTIONS:
Drug: rasagiline mesylate — 0.5 rasagiline mesylate
  Arms: Experimental 1
Drug: rasagiline mesylate 1.0 mg — 1.0 mg rasagiline mesylate
  Arms: Expermental 2

SUMMARY:
Study to look at the effectiveness, tolerability and safety of two doses of Rasagiline (0.5 mg and 1mg) in advanced Parkinson's Disease (PD) Patients who have been treated with Levodopa/Carbidopa therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have completed the Week 26 visit of TVP 1012/133 (Visit 06) in accordance with the protocol.
* Women must be postmenopausal, surgically sterile, or using adequate birth control methods. Women of childbearing potential must have a negative pregnancy test at Baseline/Month 0.
* Patients must be willing and able to give informed consent.

Exclusion Criteria:

* Serious or severe, test drug-related (probable or definite) adverse reaction in study TVP 1012/133.
* Premature discontinuation from study TVP 1012/133 for any reason.
* A clinically significant or unstable medical or surgical condition which would preclude safe and complete study participation. Such conditions may include cardiovascular, pulmonary hepatic, renal, metabolic diseases or malignancies as determined by medical history, physical exam, skin evaluation, laboratory tests, chest x-ray, or ECG.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2001-10; Primary Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
long-term safety and tolerability of rasagiline | 6 months
  To evaluate the long-term safety and tolerability of rasagiline in PD patients with motor fluctuations treated with chronic levodopa/carbidopa (LD/CD) or levodopa/benserazide (LD/BZD) therapy.

SECONDARY OUTCOMES:
long- term clinical effect of rasagiline | 6 months
  To assess the long- term clinical effect of rasagiline on the course of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Salzman, Ph.D., Study Director — Teva Neuroscience, Inc.
Locations (8):
- United States (7):
  - Margolin Brain Institute, Fresno, California
  - Emory University, Atlanta, Georgia
  - Rush - Presbyterian St. Luke's Medical Center, Chicago, Illinois
  - Creighton University, Omaha, Nebraska
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - University of Rochester, Rochester, New York
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
- CHUM-Hotel-Dieu, Montreal, Quebec, Canada